CLINICAL TRIAL: NCT01052428
Title: Molecular Mechanisms of Volume Overload-Aim 1(SCCOR in Cardiac Dysfunction and Disease)
Acronym: P1A1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Louis J. Dell'Italia, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F040601008
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Mitral Regurgitation
Keywords: Chronic MR; Volume Overload; Beta-1 receptor blocker; LV remodelling, LV dimensions; LV systolic function; LV diastolic dysfunction; Cardiac MRI
MeSH Terms: conditions — Mitral Valve Insufficiency; Edema; Ventricular Dysfunction, Left | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toprol XL (Active Comparator): beta 1 receptor blockade; generic name metoprolol succinate
  Interventions: Drug: metoprolol succinate (Toprol XL)
- Placebo (Placebo Comparator): Pill that looks like Toprol XL but does not have the active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metoprolol succinate (Toprol XL) — Toprol XL 100 mg once a day for 2 years
  Arms: Toprol XL
Drug: Placebo — Placebo 100 mg once a day for 2 years
  Arms: Placebo

SUMMARY:
The investigators hypothesize that beta-1 receptor blockade (ß1-RB) attenuates extracellular matrix (ECM) degradation and progressive adverse Left Ventricular (LV) remodeling and failure in the volume overload of mitral regurgitation (MR). Patients without coronary artery disease and moderate MR, as assessed by color/flow Doppler echocardiography, will be randomized to ß1-RB vs. placebo to address the following aims:

*Aim 1: Establish whether ß1-RB attenuates adverse LV remodeling compared to placebo in patients with non-surgical, chronic MR. Using 3-dimensional magnetic resonance imaging (MRI) and tissue tagging, LV function and geometry will be assessed at baseline and every 6 months for up to 2 years.

Aim 2: Determine whether indices of inflammation correlate with degree of LV remodeling and whether ß1-RB decrease indices of inflammation and collagen turnover. At the time of MRI, blood samples for collagen breakdown products, matrix metalloproteinase (MMP) activity, and markers of excess production of reactive inflammatory species (RIS) will be obtained and related to changes in LV remodeling defined by serial 3-dimensional MRI and tissue tagging.

DETAILED DESCRIPTION:
In Western society, the most common causes of chronic mitral regurgitation (MR) are ischemic heart disease and myxomatous degeneration of the valve, resulting in prolapse, ruptured chordae or partial flail leaflet. Current indications for surgery are only for patients with severe MR and either notable symptoms or overt Left Ventricular (LV) dysfunction (ejection fraction < 60%, end-systolic diameter > 40 mm). Therefore, despite the availability of surgery, most patients with MR of moderate severity are not immediate candidates for surgery, warranting analysis of potential beneficial effects of medical treatment. Chronic therapy with vasodilators reduces LV wall stress and thereby delays the need for valve replacement in aortic regurgitation; however, no such data are currently available in patients with chronic MR using standard vasodilators or agents that block the renin angiotensin system (RAS).

In a clinically-relevant dog model of MR, the investigators have shown increased LV ACE and chymase expression, increased LV angiotensin II but, as opposed to pressure overload, there was an absence of fibrosis with net extracellular matrix (ECM) degradation and activation of matrix metalloproteinases (MMPs). However, blockade of the RAS does not improve (and may actually exacerbate) LV remodeling in MR. Interestingly, the investigators and others have shown that ß1-receptor blockade (ß1-RB) is more effective than RAS blockade in attenuating progressive LV remodeling and ECM degradation in MR. Moreover, increased sympathetic drive and inflammation has been identified in patients with chronic MR. ß1-RB reduced plasma markers of inflammation in patients with heart failure and resulted in substantial reverse LV remodeling in patients with heart failure. Taken together, activation of the adrenergic nervous system early in the course of volume overload contributes to increased production of reactive inflammatory species (RIS) and that one mechanism underlying the salutary effects of ß1-blockade may relate to attenuation of myocardial formation of RIS with subsequent beneficial effects on MMP activation and ECM and LV remodeling and function.

ELIGIBILITY:
Inclusion Criteria:Patients who have Moderate MR documented by color flow doppler:

1. LV ejection fraction > 55%; LV end-systolic dimension < 4.0 cm.
2. Quantifiable by Doppler-Echo equal or more than moderate in severity.
3. Organic disease of the mitral valve demonstrated by echocardiography (not normal valve as in functional or ischemic MR).
4. Isolated MR (no valve disease other than mild tricuspid or pulmonic regurgitation by Doppler-Echocardiography that is often associated with mitral valve prolapse).
5. Asymptomatic (or mildly symptomatic but not considered as candidates for immediate surgery by their attending physician).

Exclusion Criteria:

1. Significant obstructive coronary artery disease and/or myocardial ischemia on graded exercise test with myocardial perfusion.
2. Previous myocardial infarction or percutaneous coronary intervention.
3. Hypertrophic cardiomyopathy, congenital or pericardial disease.
4. Aortic valve disease (> trace aortic regurgitation or mean gradient > 10 mmHg).
5. Mitral stenosis (mean gradient >5 mmHg, valve area < 1.5 cm2).
6. Intolerance or contraindication to Beta1-AR blockade.
7. Renal failure with creatinine > 2.5 mg/dl.
8. Hypertension requiring medical treatment or renal artery stenosis.
9. Severe comorbidity: liver disease, malignancy, collagen vascular, steroid requirement.
10. Pregnancy (negative pregnancy test and effective contraceptive methods are required prior to enrollment of females of childbearing potential).
11. Uncontrolled (rate > 120/min) or recent (<4 weeks) atrial fibrillation.
12. Routine, regular use of anti-inflammatory medications.

Exclusion Criteria Related to MRI

1. Severe claustrophobia.
2. Presence of a pacemaker or non-removable hearing aid.
3. Presence of metal clips in the body.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis . J. Dell'Italia, M.D, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] 1. Dell'Italia LJ. Mitral Regurgitation. In Hurst The Heart. Eds. O'Rourke, Sclhant, Alexader, Fuster. 11th Edition, Chapter 57 pp 1169-1695, 2004.
- [Background] Olson LJ, Subramanian R, Ackermann DM, Orszulak TA, Edwards WD. Surgical pathology of the mitral valve: a study of 712 cases spanning 21 years. Mayo Clin Proc. 1987 Jan;62(1):22-34. doi: 10.1016/s0025-6196(12)61522-5. PMID 3796056
- [Background] Otto CM. Timing of surgery in mitral regurgitation. Heart. 2003 Jan;89(1):100-5. doi: 10.1136/heart.89.1.100. No abstract available. PMID 12482807
- [Background] Wisenbaugh T, Essop R, Rothlisberger C, Sareli P. Effects of a single oral dose of captopril on left ventricular performance in severe mitral regurgitation. Am J Cardiol. 1992 Feb 1;69(4):348-53. doi: 10.1016/0002-9149(92)90232-n. PMID 1734647
- [Background] Rothlisberger C, Sareli P, Wisenbaugh T. Comparison of single dose nifedipine and captopril for chronic severe mitral regurgitation. Am J Cardiol. 1994 May 15;73(13):978-81. doi: 10.1016/0002-9149(94)90148-1. No abstract available. PMID 8184862
- [Background] Wisenbaugh T, Sinovich V, Dullabh A, Sareli P. Six month pilot study of captopril for mildly symptomatic, severe isolated mitral and isolated aortic regurgitation. J Heart Valve Dis. 1994 Mar;3(2):197-204. PMID 8012639
- [Background] Marcotte F, Honos GN, Walling AD, Beauvais D, Blais MJ, Daoust C, Lisbona A, McCans JL. Effect of angiotensin-converting enzyme inhibitor therapy in mitral regurgitation with normal left ventricular function. Can J Cardiol. 1997 May;13(5):479-85. PMID 9179087
- [Background] Host U, Kelbaek H, Hildebrandt P, Skagen K, Aldershvile J. Effect of ramipril on mitral regurgitation secondary to mitral valve prolapse. Am J Cardiol. 1997 Sep 1;80(5):655-8. doi: 10.1016/s0002-9149(97)00445-1. PMID 9295005
- [Background] Tischler MD, Rowan M, LeWinter MM. Effect of enalapril therapy on left ventricular mass and volumes in asymptomatic chronic, severe mitral regurgitation secondary to mitral valve prolapse. Am J Cardiol. 1998 Jul 15;82(2):242-5. doi: 10.1016/s0002-9149(98)00325-7. PMID 9678300
- [Background] Dujardin KS, Enriquez-Sarano M, Bailey KR, Seward JB, Tajik AJ. Effect of losartan on degree of mitral regurgitation quantified by echocardiography. Am J Cardiol. 2001 Mar 1;87(5):570-6. doi: 10.1016/s0002-9149(00)01433-8. PMID 11230841
- [Background] Gaasch WH, Aurigemma GP. Inhibition of the renin-angiotensin system and the left ventricular adaptation to mitral regurgitation. J Am Coll Cardiol. 2002 Apr 17;39(8):1380-3. doi: 10.1016/s0735-1097(02)01766-7. No abstract available. PMID 11955859
- [Background] Stewart JA Jr, Wei CC, Brower GL, Rynders PE, Hankes GH, Dillon AR, Lucchesi PA, Janicki JS, Dell'Italia LJ. Cardiac mast cell- and chymase-mediated matrix metalloproteinase activity and left ventricular remodeling in mitral regurgitation in the dog. J Mol Cell Cardiol. 2003 Mar;35(3):311-9. doi: 10.1016/s0022-2828(03)00013-0. PMID 12676546
- [Background] Perry GJ, Wei CC, Hankes GH, Dillon SR, Rynders P, Mukherjee R, Spinale FG, Dell'Italia LJ. Angiotensin II receptor blockade does not improve left ventricular function and remodeling in subacute mitral regurgitation in the dog. J Am Coll Cardiol. 2002 Apr 17;39(8):1374-9. doi: 10.1016/s0735-1097(02)01763-1. PMID 11955858
- [Background] Dell'italia LJ, Balcells E, Meng QC, Su X, Schultz D, Bishop SP, Machida N, Straeter-Knowlen IM, Hankes GH, Dillon R, Cartee RE, Oparil S. Volume-overload cardiac hypertrophy is unaffected by ACE inhibitor treatment in dogs. Am J Physiol. 1997 Aug;273(2 Pt 2):H961-70. doi: 10.1152/ajpheart.1997.273.2.H961. PMID 9277516
- [Background] Nemoto S, Hamawaki M, De Freitas G, Carabello BA. Differential effects of the angiotensin-converting enzyme inhibitor lisinopril versus the beta-adrenergic receptor blocker atenolol on hemodynamics and left ventricular contractile function in experimental mitral regurgitation. J Am Coll Cardiol. 2002 Jul 3;40(1):149-54. doi: 10.1016/s0735-1097(02)01926-5. PMID 12103269
- [Background] Tallaj J, Wei CC, Hankes GH, Holland M, Rynders P, Dillon AR, Ardell JL, Armour JA, Lucchesi PA, Dell'Italia LJ. Beta1-adrenergic receptor blockade attenuates angiotensin II-mediated catecholamine release into the cardiac interstitium in mitral regurgitation. Circulation. 2003 Jul 15;108(2):225-30. doi: 10.1161/01.CIR.0000079226.48637.5A. Epub 2003 Jul 7. PMID 12847066
- [Background] Tsutsui H, Spinale FG, Nagatsu M, Schmid PG, Ishihara K, DeFreyte G, Cooper G 4th, Carabello BA. Effects of chronic beta-adrenergic blockade on the left ventricular and cardiocyte abnormalities of chronic canine mitral regurgitation. J Clin Invest. 1994 Jun;93(6):2639-48. doi: 10.1172/JCI117277. PMID 7911128
- [Background] Mehta RH, Supiano MA, Oral H, Grossman PM, Montgomery DS, Smith MJ, Starling MR. Compared with control subjects, the systemic sympathetic nervous system is activated in patients with mitral regurgitation. Am Heart J. 2003 Jun;145(6):1078-85. doi: 10.1016/S0002-8703(03)00111-X. PMID 12796766
- [Background] Mehta RH, Supiano MA, Oral H, Grossman PM, Petrusha JA, Montgomery DG, Briesmiester KA, Smith MJ, Starling MR. Relation of systemic sympathetic nervous system activation to echocardiographic left ventricular size and performance and its implications in patients with mitral regurgitation. Am J Cardiol. 2000 Dec 1;86(11):1193-7. doi: 10.1016/s0002-9149(00)01201-7. PMID 11090790
- [Background] Oral H, Sivasubramanian N, Dyke DB, Mehta RH, Grossman PM, Briesmiester K, Fay WP, Pagani FD, Bolling SF, Mann DL, Starling MR. Myocardial proinflammatory cytokine expression and left ventricular remodeling in patients with chronic mitral regurgitation. Circulation. 2003 Feb 18;107(6):831-7. doi: 10.1161/01.cir.0000049745.38594.6d. PMID 12591752
- [Background] Kukin ML, Kalman J, Charney RH, Levy DK, Buchholz-Varley C, Ocampo ON, Eng C. Prospective, randomized comparison of effect of long-term treatment with metoprolol or carvedilol on symptoms, exercise, ejection fraction, and oxidative stress in heart failure. Circulation. 1999 May 25;99(20):2645-51. doi: 10.1161/01.cir.99.20.2645. PMID 10338457
- [Background] Yue TL, Cheng HY, Lysko PG, McKenna PJ, Feuerstein R, Gu JL, Lysko KA, Davis LL, Feuerstein G. Carvedilol, a new vasodilator and beta adrenoceptor antagonist, is an antioxidant and free radical scavenger. J Pharmacol Exp Ther. 1992 Oct;263(1):92-8. PMID 1357162
- [Background] Flesch M, Maack C, Cremers B, Baumer AT, Sudkamp M, Bohm M. Effect of beta-blockers on free radical-induced cardiac contractile dysfunction. Circulation. 1999 Jul 27;100(4):346-53. doi: 10.1161/01.cir.100.4.346. PMID 10421593
- [Background] Chin BS, Langford NJ, Nuttall SL, Gibbs CR, Blann AD, Lip GY. Anti-oxidative properties of beta-blockers and angiotensin-converting enzyme inhibitors in congestive heart failure. Eur J Heart Fail. 2003 Mar;5(2):171-4. doi: 10.1016/s1388-9842(02)00251-9. PMID 12644008
- [Background] Bristow MR. Mechanistic and clinical rationales for using beta-blockers in heart failure. J Card Fail. 2000 Jun;6(2 Suppl 1):8-14. PMID 10908093
- [Background] Diez J, Querejeta R, Lopez B, Gonzalez A, Larman M, Martinez Ubago JL. Losartan-dependent regression of myocardial fibrosis is associated with reduction of left ventricular chamber stiffness in hypertensive patients. Circulation. 2002 May 28;105(21):2512-7. doi: 10.1161/01.cir.0000017264.66561.3d. PMID 12034658
- [Background] Querejeta R, Varo N, Lopez B, Larman M, Artinano E, Etayo JC, Martinez Ubago JL, Gutierrez-Stampa M, Emparanza JI, Gil MJ, Monreal I, Mindan JP, Diez J. Serum carboxy-terminal propeptide of procollagen type I is a marker of myocardial fibrosis in hypertensive heart disease. Circulation. 2000 Apr 11;101(14):1729-35. doi: 10.1161/01.cir.101.14.1729. PMID 10758057
- [Background] Lopez B, Querejeta R, Varo N, Gonzalez A, Larman M, Martinez Ubago JL, Diez J. Usefulness of serum carboxy-terminal propeptide of procollagen type I in assessment of the cardioreparative ability of antihypertensive treatment in hypertensive patients. Circulation. 2001 Jul 17;104(3):286-91. doi: 10.1161/01.cir.104.3.286. PMID 11457746
- [Background] Cracowski JL, Tremel F, Marpeau C, Baguet JP, Stanke-Labesque F, Mallion JM, Bessard G. Increased formation of F(2)-isoprostanes in patients with severe heart failure. Heart. 2000 Oct;84(4):439-40. doi: 10.1136/heart.84.4.439. No abstract available. PMID 10995421
- [Background] Mallat Z, Philip I, Lebret M, Chatel D, Maclouf J, Tedgui A. Elevated levels of 8-iso-prostaglandin F2alpha in pericardial fluid of patients with heart failure: a potential role for in vivo oxidant stress in ventricular dilatation and progression to heart failure. Circulation. 1998 Apr 28;97(16):1536-9. doi: 10.1161/01.cir.97.16.1536. PMID 9593557
- [Background] Nonaka-Sarukawa M, Yamamoto K, Aoki H, Takano H, Katsuki T, Ikeda U, Shimada K. Increased urinary 15-F2t-isoprostane concentrations in patients with non-ischaemic congestive heart failure: a marker of oxidative stress. Heart. 2003 Aug;89(8):871-4. doi: 10.1136/heart.89.8.871. PMID 12860861
- [Background] Mak S, Newton GE. The oxidative stress hypothesis of congestive heart failure: radical thoughts. Chest. 2001 Dec;120(6):2035-46. doi: 10.1378/chest.120.6.2035. PMID 11742938
- [Background] Rouleau JL, Pitt B, Dhalla NS, Dhalla KS, Swedberg K, Hansen MS, Stanton E, Lapointe N, Packer M; Canadian Prospective RandOmized FlosequInan Longevity Evaluation Investigators. Prognostic importance of the oxidized product of catecholamines, adrenolutin, in patients with severe heart failure. Am Heart J. 2003 May;145(5):926-32. doi: 10.1016/s0002-8703(02)94782-4. PMID 12766756
- [Background] Lopez Farre A, Casado S. Heart failure, redox alterations, and endothelial dysfunction. Hypertension. 2001 Dec 1;38(6):1400-5. doi: 10.1161/hy1201.099612. PMID 11751725
- [Background] Sorescu D, Griendling KK. Reactive oxygen species, mitochondria, and NAD(P)H oxidases in the development and progression of heart failure. Congest Heart Fail. 2002 May-Jun;8(3):132-40. doi: 10.1111/j.1527-5299.2002.00717.x. PMID 12045381
- [Background] Wachtell K, Palmieri V, Olsen MH, Gerdts E, Papademetriou V, Nieminen MS, Smith G, Dahlof B, Aurigemma GP, Devereux RB. Change in systolic left ventricular performance after 3 years of antihypertensive treatment: the Losartan Intervention for Endpoint (LIFE) Study. Circulation. 2002 Jul 9;106(2):227-32. doi: 10.1161/01.cir.0000021601.49664.2a. PMID 12105163
- [Derived] Ahmed MI, Aban I, Lloyd SG, Gupta H, Howard G, Inusah S, Peri K, Robinson J, Smith P, McGiffin DC, Schiros CG, Denney T Jr, Dell'Italia LJ. A randomized controlled phase IIb trial of beta(1)-receptor blockade for chronic degenerative mitral regurgitation. J Am Coll Cardiol. 2012 Aug 28;60(9):833-8. doi: 10.1016/j.jacc.2012.04.029. Epub 2012 Jul 18. PMID 22818065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Toprol-XL
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Toprol-XL | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 0 | 3 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.3) | 55.9 (9.2) | 54.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular End Diastolic Volume Indexed to Body Surface Area
Description: Left Ventricular End Diastolic Volume Indexed to Body Surface Area: As an indicator of heart size, the blood volume of the heart is related to the body size. The end diastolic volume is the blood volume of the heart at the end of filling, just before contraction. The relation of heart blood volume to body size is more accurate in determining pathology because larger people require a larger heart blood volume. The values that are too high or too low indicate a diseased myocardium.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: ml/m^2
Groups:
- Toprol XL: Generic name metoprolol succinate
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
ml/m^2
  Month 0 (n=19,19) | 91.66 (16.48) | 95.74 (19.89)
  Month 3 (n=1,0) | 90.93 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 90.84 (16.39) | 95.24 (18.52)
  Month 9 (n=1,0) | 70.56 (NA) — n=1 | NA (NA) — no observation
  Month 12 (n=14,15) | 88.99 (16.63) | 95.71 (20.59)
  Month 15 (n=3,2) | 82.73 (14.18) | 98.16 (2.89)
  Month 18 (n=14,18) | 90.16 (21.49) | 97.6 (19.82)
  Month 21 (n=5,0) | 85.75 (15.24) | NA (NA) — no observation
  Month 24 (n=16,18) | 87.31 (20.91) | 95.16 (23.94)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; The differences in the rate of progression of the outcome measures were the focus of the comparisons over time between the treatment groups. A significant interaction effect between time and treatment group in the mixed model is the measure of treatment effect. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes and the number of Participants for each interval is indicated as (n=x,y); Test type: Superiority or Other; p = 0.4568, Mixed Models Analysis

2. Primary Outcome: Left Ventricular End-diastolic Mass Indexed to Left Ventricular End-diastolic Volume
Description: Left Ventricular End-diastolic Mass Indexed to Left Ventricular End-diastolic Volume As an indicator of heart muscle mass and heart blood volume, the mass indexed to end diastolic volume determines whether there is an adequate amount of heart muscle to pump the heart blood volume obtained from a three-dimensional analysis. The values that are too high or too low indicate a diseased myocardium.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: g/ml
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
g/ml
  Month 0 (n=19,19) | 0.61 (0.13) | 0.61 (0.12)
  Month 3 (n=1,0) | 0.53 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 0.62 (0.11) | 0.6 (0.12)
  Month 9 (n=1,1) | 0.67 (NA) — n=1 | 0.53 (NA) — n=1
  Month 12 (n=14,15) | 0.65 (0.12) | 0.60 (0.1)
  Month 15 (n=3,2) | 0.65 (0.18) | 0.55 (0.05)
  Month 18 (n=14,18) | 0.65 (0.11) | 0.59 (0.09)
  Month 21 (n=5,0) | 0.61 (0.13) | NA (NA) — no observation
  Month 24 (n=16,18) | 0.64 (0.12) | 0.62 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1967, Mixed Models Analysis — not adjusted for multiple comparisons

3. Primary Outcome: Left Ventricular End-Diastolic Radius to Wall Thickness
Description: Left Ventricular End-Diastolic Radius to Wall Thickness As an indicator of heart muscle mass and heart volume chamber diameter, the end-diastolic radius indexed to end diastolic wall thickness determines whether there is an adequate amount of heart muscle to pump the heart blood volume obtained from a two-dimensional analysis. The values that are too high or too low indicate a diseased myocardium.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
unitless
  Month 0 (n=19,19) | 4.76 (0.92) | 4.69 (0.92)
  Month 3 (n=1,0) | 5.02 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 4.51 (0.62) | 4.85 (0.92)
  Month 9 (n=1,1) | 4.15 (NA) — n=1 | 5.74 (NA) — n=1
  Month 12 (n=14,15) | 4.46 (0.64) | 4.79 (0.95)
  Month 15 (n=3,2) | 4.61 (1.69) | 5.02 (0.48)
  Month 18 (n=14,18) | 4.43 (0.69) | 4.77 (0.83)
  Month 21 (n=5,0) | 4.72 (0.91) | NA (NA) — no observation
  Month 24 (n=16,18) | 4.52 (0.78) | 4.59 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — not adjusted for multiple comparisons

4. Primary Outcome: Left Ventricular End Systolic Volume Indexed to Body Surface Area
Description: Left Ventricular End Systolic Volume Indexed to Body Surface Area As an indicator of heart size, the blood volume of the heart is related to the body size. The end systolic volume is the blood volume of the heart at the end of contraction and is an index of the pump function of the heart. This relation to body size is more accurate in determining pathology because larger people require a larger heart blood volume. The values that are too high or too low indicate a diseased myocardium.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
ml/m^2
  Month 0 (n=19,19) | 34.01 (6.86) | 35.98 (8.12)
  Month 3 (n=1,0) | 32.83 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 32.53 (6.15) | 36.53 (6.76)
  Month 9 (n=1,0) | 40.99 (NA) — n=1 | NA (NA) — no observation
  Month 12 (n=14,15) | 33.70 (7.62) | 35.89 (10.52)
  Month 15 (n=3,2) | 47.25 (21.32) | 30.97 (2.9)
  Month 18 (n=14,18) | 34.99 (10.08) | 36.72 (8.04)
  Month 21 (n=5,0) | 39.97 (13.22) | NA (NA) — no observation
  Month 24 (n=16,18) | 34.47 (8.72) | 35.13 (10.47)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis — not adjusted for multiple comparisons

5. Primary Outcome: Left Ventricular Ejection Fraction
Description: Left Ventricular Ejection Fraction Is a calculation of heart pump function determined from the volume after complete filling minus the volume after complete contraction divided by the volume after complete filling. A value of 55% or greater is normal.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
percent
  Month 0 (n=19,19) | 62.62 (5.25) | 62.09 (6.45)
  Month 3 (n=1,0) | 63.90 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 63.80 (6.15) | 61.29 (4.66)
  Month 9 (n=1,1) | 41.90 (NA) — n=1 | 54.81 (NA) — n=1
  Month 12 (n=14,15) | 61.70 (6.87) | 62.77 (6.14)
  Month 15 (n=3,2) | 44.70 (16.03) | 68.47 (2.02)
  Month 18 (n=14,18) | 60.95 (8.23) | 62.05 (5.68)
  Month 21 (n=5,0) | 53.79 (11.20) | NA (NA) — no observation
  Month 24 (n=16,18) | 59.95 (8.27) | 63.02 (6.05)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — not adjusted for multiple comparisons

6. Primary Outcome: Systolic Longitudinal Strain
Description: Systolic Longitudinal Strain. By identifying two points on the heart, the strain is the difference between the distance between these two points at the end of filling of the heart and the end of contraction divided by the length at the end of filling. Thus, the measure is like the ejection fraction, however the strain is more localized to a specified segment in the heart muscle. The higher values indicate a healthy heart.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: percent/%Systolic interval
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
percent/%Systolic interval
  Month 0 (n=19,19) | 87.94 (27.44) | 82.55 (29.31)
  Month 3 (n=1,0) | 115.07 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 45.90 (34.56) | 78.68 (22.97)
  Month 9 (n=1,0) | 37.2 (NA) — n=1 | NA (NA) — no observation
  Month 12 (n=14,15) | 87.85 (26.07) | 80.04 (20.58)
  Month 15 (n=3,2) | 52.95 (20.87) | 88.34 (6.70)
  Month 18 (n=14,18) | 88.11 (34.96) | 79.29 (22.14)
  Month 21 (n=5,0) | 67.53 (26.81) | NA (NA) — no observation
  Month 24 (n=16,18) | 79.94 (24.24) | 85.18 (32.2)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis — not adjusted for multiple comparisons

7. Primary Outcome: Peak Early Filling Rate: Rate of Change Over Time
Description: Peak Early Filling Rate The peak early filling rate of change is calculated from the slope of the volume during the early filling of the heart with respect to time. The higher values indicate a very healthy heart muscle and lower values are indicative of a very stiff muscle.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: EDV/sec
Arm/Group | Placebo | Toprol XL
Number analyzed (Participants) | 19 | 19
EDV/sec
  Month 0 (n=19,19) | 2.27 (0.61) | 2.12 (0.57)
  Month 3 (n=1,0) | 2.58 (NA) — n=1 | NA (NA) — no observation
  Month 6 (n=17,19) | 2.38 (0.53) | 2.08 (0.55)
  Month 9 (n=1,0) | 1.56 (NA) — n=1 | NA (NA) — no observation
  Month 12 (n=14,15) | 2.26 (0.52) | 2.24 (0.46)
  Month 15 (n=3,2) | 1.83 (1.56) | 2.28 (0.47)
  Month 18 (n=14,18) | 1.95 (0.63) | 2.26 (0.56)
  Month 21 (n=5,0) | 1.73 (0.99) | NA (NA) — no observation
  Month 24 (n=16,18) | 2.17 (0.60) | 2.25 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Toprol XL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 2 years
Description: visit is every 6 months
Arm/Group | Placebo | Toprol-XL
Serious Adverse Events (participants affected / at risk) | 7/19 | 4/19
Other Adverse Events (participants affected / at risk) | 6/19 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Toprol-XL (N=19)
Continued right calf pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Death (Surgical and medical procedures) | 0 (0) | 1 (1) — Death due to bloodclot two weeks after liposuction
Hearing loss and tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Mitral Valve Replacement (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve repair (Cardiac disorders) | 5 (5) | 2 (2)
Pleural effusion and thoracentesis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prostrate cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Toprol-XL (N=19)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
colon polyp removed (Gastrointestinal disorders) | 0 (0) | 1 (1)
headaches (Nervous system disorders) | 1 (1) | 0 (0)
hyperlipidemia (Endocrine disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
left foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
left upper arm broken (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nodule rt of thyroid (Endocrine disorders) | 1 (1) | 0 (0)
sinus infection (Infections and infestations) | 0 (0) | 1 (1)
tendonitis rt shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No